CLINICAL TRIAL: NCT02725619
Title: Neural Mechanisms of CBT for Anxiety in Children With Autism: Randomized Controlled Trial
Brief Title: CBT for Anxiety in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1211011144B; 1R01HD083881-01A1 (NIH)
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Experimental): CBT is dedicated to developing coping skills for managing anxiety such as emotion regulation and cognitive reappraisal. Children first learn and practice these skills during one-on-one, weekly sessions with experienced therapists and then apply this skills to navigate anxiety-producing situations as home, school and community. A key component of CBT involves exposure exercises, facing feared situations repeatedly while using the emotion regulation skills and remaining in the situations until anxiety is substantially reduced or become easy to tolerate. The feared situations are ordered from least to most distressing during therapy sessions in collaboration with the child and their parent. The unique combination of anxiety and ASD symptoms of social impairment and restricted/repetitive behavior is addressed in dedicated child and parent modules.
  Interventions: Behavioral: CBT
- Psychoeducation and Supportive Therapy (PST) (Active Comparator): Psychoeducation and Supportive Therapy includes learning about and discussing issues of diagnosis, treatment and educational services can also benefit children with ASD and their families. Each PST session starts with a review of events of the past week and include queries of topics such as school, interests, and family with an overarching goal of enhancing subjective well-being. The clinician, through the use of supportive, empathic and nondirective actions, will provide the participant with a "sounding-board" so that they can voice their concerns regarding specific problems that may require discussion and assistance. A major objective is to provide a clinical contact that enables participants to think through and discuss their concerns with a sympathetic adult. Subjects randomized to PST will be offered CBT after completion of the endpoint assessments.
  Interventions: Behavioral: PST

INTERVENTIONS:
Behavioral: CBT
  Other Names: Behavior therapy
  Arms: Cognitive-Behavioral Therapy (CBT)
Behavioral: PST
  Other Names: Supportive psychotherapy
  Arms: Psychoeducation and Supportive Therapy (PST)

SUMMARY:
This is a randomized controlled trial of Cognitive Behavioral Therapy (CBT) versus Psychoeducation and Supportive Therapy (PST) in children with Autism Spectrum Disorder and moderate to severe anxiety. The study will utilize fMRI to identify CBT-invoked changes in levels of activity/functional connectivity within the neural circuits involved in emotion regulation and social perception. Matched typically developing children without autism and/or anxiety will be scanned twice, 16 weeks apart, to enable interpretation of treatment-evoked change relative to normative development.

DETAILED DESCRIPTION:
Anxiety is among the most common concerns in children with autism spectrum disorder (ASD) who seek mental health services, causing suffering and family stress and exacerbating social disability. Cognitive-Behavioral Therapy (CBT) is a promising treatment for anxiety in children with high-functioning ASD, but the neural mechanisms supporting response to this treatment have not been studied. The neural-systems-level targets of CBT for anxiety in children with ASD will be investigated by evaluating brain indices of socio-emotional functioning with functional magnetic resonance imaging (fMRI) before and after treatment. CBT teaches emotion regulation skills, such as cognitive reappraisal, followed by behavioral exposure to anxiety-provoking situations. It is hypothesized that CBT aimed at the reduction of anxiety will enhance the neural circuitry that subserves the experience and regulation of emotions. This is a randomized controlled trial of CBT vs. Psychoeducation and Supportive Therapy (PST) in 100 school-age children with high-functioning ASD and moderate to severe anxiety. In addition, 50 matched typically-developing (TD) children will be scanned twice with a 16-week interval to enable interpretation of change in brain function in children with ASD after CBT vs. PST relative to TD children. CBT for anxiety will be provided using a structured manual that has been modified for children with ASD by increasing parental participation and addressing the role of core ASD symptoms in the experience and expression of anxiety. Subjects will be comprehensively characterized with regard to ASD diagnosis, IQ, adaptive behavior, and comorbid psychopathology. Functional MRI will be collected as the subjects perform tasks involving emotion regulation, emotional face perception, biological motion perception, and resting state.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls, ages 8 to 14 inclusive
* Diagnosis of autism spectrum disorder
* Diagnosis of anxiety disorder and clinically significant level of anxiety
* Full scale IQ and Verbal IQ > 70
* Unmedicated or on stable medication with no planned changes for duration of study
* able to meet MRI safety (e.g., no metal medical implants) and data quality requirements (e.g., able to keep head still during scanning)

Exclusion Criteria:

* Presence of a known serious medical condition that would interfere with participation in the study
* Present of a current psychiatric disorder that requires immediate clinical attention
* A previous adequate trial of CBT for anxiety within the past 2 years.

Note: This study will also recruit healthy volunteers (typically developing children without past or current mental health concerns).

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2016-04; Primary Completion 2022-04-05 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | change from baseline (week 0) at midpoint (week 8)
  The PARS is a 50-item semi-structures interview of anxiety that will be conducted by an expert clinician. Endorsed symptoms are rated using 0-5 severity scale on 7 dimensions and a sum of scores for 5 of 7 dimensions constitute the total PARS score.
Pediatric Anxiety Rating Scale (PARS) | change from baseline (week 0) at endpoint (week 16)
  The PARS is a 50-item semi-structures interview of anxiety that will be conducted by an expert clinician. Endorsed symptoms are rated using 0-5 severity scale on 7 dimensions and a sum of scores for 5 of 7 dimensions constitute the total PARS score.
Clinical Global Impression - Improvement (CGI-I) scale | change from baseline (week 0) at midpoint (week 8)
  The CGI-I reflects the IE's assessment of overall change of the target symptoms from baseline on a scale from very much improved (score of 1) through no change (score of 4) to very much worse (score of 7). By convention, ratings of very much improved (score of 1) and much improved (score of 2) define positive response.
Clinical Global Impression - Improvement (CGI-I) scale | change from baseline (week 0) at endpoint (week 16)
  The CGI-I reflects the IE's assessment of overall change of the target symptoms from baseline on a scale from very much improved (score of 1) through no change (score of 4) to very much worse (score of 7). By convention, ratings of very much improved (score of 1) and much improved (score of 2) define positive response.
blood oxygenation level dependent signal (BOLD) during down-regulation versus passive viewing of affective images. | change from baseline (week 0) at endpoint (week 16)
  During a Functional Magnetic Resonance Imaging (fMRI), subjects will view neutral and affect-inducing pictures selected to be appropriate for children. During the emotion regulation task, subjects are asked to either simply look at the pictures or to down-regulate their emotional reaction to the picture.

SECONDARY OUTCOMES:
blood oxygenation level dependent signal (BOLD) during emotional face perception task | change from baseline (week 0) at endpoint (week 16)
  During a Functional Magnetic Resonance Imaging (fMRI), subjects will complete the emotional face perception task. This task involves subjects being asked to view and match emotional faces and geometrical shapes. During "match emotion" blocks, participants view a trio of angry, fearful, or neutral faces and match emotional expression of one of two faces to the target face.

OTHER OUTCOMES:
blood oxygenation level dependent signal (BOLD) during perception of biological versus scrambled motion. | change from baseline (week 0) at endpoint (week 16)
  During a Functional Magnetic Resonance Imaging (fMRI), participants will perform the biological motion perception task. This task involves viewing coherent and scrambled point-light displays of biological motion created from motion capture data. The coherent motion displays feature an adult performing easily recognizable movements, such as playing pat-a-cake. The scrambled motion animations were created by randomly selecting 16 points from the biological motion displays and plotting their trajectories on a black background.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All data generated by this study will be delivered to the National Database for Autism Research (NDAR) as required.

REFERENCES:
- [Result] Sukhodolsky DG, Bloch MH, Panza KE, Reichow B. Cognitive-behavioral therapy for anxiety in children with high-functioning autism: a meta-analysis. Pediatrics. 2013 Nov;132(5):e1341-50. doi: 10.1542/peds.2013-1193. Epub 2013 Oct 28. PMID 24167175
- [Result] Sukhodolsky DG, Scahill L, Gadow KD, Arnold LE, Aman MG, McDougle CJ, McCracken JT, Tierney E, Williams White S, Lecavalier L, Vitiello B. Parent-rated anxiety symptoms in children with pervasive developmental disorders: frequency and association with core autism symptoms and cognitive functioning. J Abnorm Child Psychol. 2008 Jan;36(1):117-28. doi: 10.1007/s10802-007-9165-9. Epub 2007 Aug 3. PMID 17674186